CLINICAL TRIAL: NCT07048496
Title: Intravesical Treatment of Bladder Cancer at Home, Multi-modal Treatment Support
Acronym: BCG at Home
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Daniel Lee, MD, MS, Principal Investigator, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 853376; UPCC 04823 (Other: ACC)
Record Dates: First submitted 2025-05-06; First posted 2025-07-02 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: BCG delivery at home — The BCG at home project will be a single-arm prospective pilot, to evaluate the feasibility, scalability and effectiveness of home treatment, and utilize the BB-Bot (chatbot) for PRO and adverse event measurement.

SUMMARY:
The proposed project will have two separate cohorts. The first will be to perform a more in-depth qualitative assessment of the barriers and facilitators for treatment compliance for non-muscle invasive bladder cancer. The second arm will be to create and test a BCG at home program. Participants in the second cohort will be enrolled in a conversational agent to measure patient symptoms and quality of life and improve self-efficacy.

DETAILED DESCRIPTION:
The proposed project will have two separate cohorts. The first will be to perform a more in-depth qualitative assessment of the barriers and facilitators for treatment compliance for non-muscle invasive bladder cancer. The second arm will be to create and test a BCG at home program. Participants in the second cohort will be enrolled in a conversational agent to measure patient symptoms and quality of life and improve self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients in Cohort 1

* Age 18 years or older;
* completed intravesical treatment for non-muscle invasive bladder cancer within the past year Cohort 1 inclusion criteria for key stakeholders
* Age 18 years or older;
* experience with the delivery of BCG delivery for more than 2 years

Cohort 2 inclusion criteria

* Age 18 years or older;
* diagnosed with non-muscle invasive bladder cancer and prescribed BCG for initial therapy

Exclusion Criteria:

Cohort 1 exclusion criteria

• inability to provide informed consent

Cohort 2 exclusion criteria

* inability to provide informed consent
* inability to undergo catheterization (i.e. - history of urethral stricture)
* inability to receive BCG therapy (i.e. - previous reaction with BCG)
* no access to mobile phone
* inability to respond to written conversations in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-05 (Actual); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence to BCG therapy at 3 months after study initiation | 3 months after study initiation
  The primary outcome will be the rate of adherence to AUA guidelines for BCG therapy as measured by successful treatments of BCG compared to expected treatments. For each participant, adherence will be calculated both as the percentage of adherent doses, evaluable for study participants

SECONDARY OUTCOMES:
• Self efficacy as measured by the validated General Self efficacy scale, a 10-item scale, measured at 3 months after study initiation | 3 months after study initiation
  The secondary outcomes will include self-efficacy and symptom management.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No